CLINICAL TRIAL: NCT00006489
Title: Naltrexone and Cognitive-Behavioral Therapy for Patients With Alcoholism and Post-Traumatic Stress Disorder
Brief Title: Treatment for Alcoholism and Post-Traumatic Stress Disorder (Naltrexone)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: NIAAAFOA12428; R01AA012428 (NIH); NIH grant R01-AA-012428
Record Dates: First submitted 2000-11-08; First posted 2000-11-09 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-03

CONDITIONS: Alcoholism; Alcohol Dependence; Post-Traumatic Stress Disorder
Keywords: Alcoholism; Alcohol Dependence; Post-Traumatic Stress Disorder; Naltrexone; Cognitive Behavior Therapy
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic | interventions — Cognitive Behavioral Therapy; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Naltrexone alone (Active Comparator): Naltrexone alone
  Interventions: Drug: Naltrexone
- Naltrexone with CBT for PTSD (Active Comparator): Naltrexone with CBT for PTSD
  Interventions: Behavioral: Cognitive-Behavioral Therapy; Drug: Naltrexone
- Placebo with CBT for PTSD (Active Comparator): Placebo with CBT for PTSD
  Interventions: Behavioral: Cognitive-Behavioral Therapy
- Placebo alone (Placebo Comparator): Placebo alone
  Interventions: Drug: Placebo

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy — Twelve weekly 90-minute individual therapy sessions followed by (6) 90-minute sessions every other week
  Arms: Naltrexone with CBT for PTSD; Placebo with CBT for PTSD
Drug: Naltrexone — Daily dosing 100 mg for 24 weeks
  Arms: Naltrexone alone; Naltrexone with CBT for PTSD
Drug: Placebo — Pill Placebo daily dosing 24 weeks
  Arms: Placebo alone

SUMMARY:
This study will evaluate naltrexone and cognitive-behavioral therapy treatments for alcohol dependence and post-traumatic stress disorder (PTSD). Subjects will be randomly assigned a 6-month treatment of either: 1) naltrexone alone, 2) naltrexone with PTSD psychosocial therapy, 3) a placebo with PTSD psychosocial therapy, or 4) placebo alone. An enhanced medication management intervention will accompany all treatment conditions. Follow-up assessments will be completed at 9 and 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for alcohol dependence and post-traumatic stress disorder.
* Heavy drinking in the past 30 days (an average of more than 12 alcohol drinks per week with at least 1 day of 4 or more drinks).
* Successfully complete medical detoxification.
* Exhibit clinically significant trauma-related symptoms.
* Live in a commutable distance to the University of Pennsylvania and agree to follow-up visits.
* Aged between 18 and 65 years old.
* Able to provide an informed consent.
* Speak and read English.

Exclusion Criteria:

* Current diagnosis of any substance dependence other than alcohol, nicotine, or cannabis.
* Evidence of opiate use in the past 30 days.
* Significant risk of violence or history of serious violent behavior during the past year.
* Continued contact with an intimate partner if assault by the partner is the index trauma.
* Changes in dosage or medication for any SSRI treatment in the three months prior to entering the study.
* Unstable or serious medical illness.
* Current severe psychiatric symptom.
* Mental retardation or another pervasive developmental disorder.
* Use of an investigational medication in the past 30 days.
* Pregnant, nursing or not using reliable contraception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2000-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edna B. Foa, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Center for Anxiety, University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Zang Y, Yu J, Chazin D, Asnaani A, Zandberg LJ, Foa EB. Changes in coping behavior in a randomized controlled trial of concurrent treatment for PTSD and alcohol dependence. Behav Res Ther. 2017 Mar;90:9-15. doi: 10.1016/j.brat.2016.11.013. Epub 2016 Nov 24. PMID 27930926
- [Derived] Kaczkurkin AN, Asnaani A, Alpert E, Foa EB. The impact of treatment condition and the lagged effects of PTSD symptom severity and alcohol use on changes in alcohol craving. Behav Res Ther. 2016 Apr;79:7-14. doi: 10.1016/j.brat.2016.02.001. Epub 2016 Feb 15. PMID 26905901
- [Derived] Foa EB, Yusko DA, McLean CP, Suvak MK, Bux DA Jr, Oslin D, O'Brien CP, Imms P, Riggs DS, Volpicelli J. Concurrent naltrexone and prolonged exposure therapy for patients with comorbid alcohol dependence and PTSD: a randomized clinical trial. JAMA. 2013 Aug 7;310(5):488-95. doi: 10.1001/jama.2013.8268. PMID 23925619
- [Derived] Powers MB, Gillihan SJ, Rosenfield D, Jerud AB, Foa EB. Reliability and validity of the PDS and PSS-I among participants with PTSD and alcohol dependence. J Anxiety Disord. 2012 Jun;26(5):617-23. doi: 10.1016/j.janxdis.2012.02.013. Epub 2012 Mar 3. PMID 22480715

RESULTS

PARTICIPANT FLOW:
Groups:
- Naltrexone + Supportive Counseling: Naltrexone alone
  Naltrexone: Daily dosing 100 mg for 24 weeks
- Naltrexone + CBT (Prolonged Exposure Therapy): Naltrexone with CBT for PTSD
  Cognitive-Behavioral Therapy: Twelve weekly 90-minute individual therapy sessions followed by (6) 90-minute sessions every other week
  Naltrexone: Daily dosing 100 mg for 24 weeks
- Placebo + CBT (Prolonged Exposure Therapy): Placebo with CBT for PTSD
  Cognitive-Behavioral Therapy: Twelve weekly 90-minute individual therapy sessions followed by (6) 90-minute sessions every other week
- Placebo + Supportive Counseling: Placebo alone
  Placebo: Pill Placebo daily dosing 24 weeks
Period: Overall Study
Arm/Group | Naltrexone + Supportive Counseling | Naltrexone + CBT (Prolonged Exposure Therapy) | Placebo + CBT (Prolonged Exposure Therapy) | Placebo + Supportive Counseling
Started | 42 | 40 | 40 | 43
Completed | 29 | 26 | 25 | 32
Not Completed | 13 | 14 | 15 | 11
Not completed — Adverse Event | 3 | 2 | 4 | 3
Not completed — Withdrawal by Subject | 10 | 9 | 9 | 6
Not completed — Scheduling Conflict | 0 | 3 | 2 | 1
Not completed — Death | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone + Supportive Counseling | Naltrexone + CBT (Prolonged Exposure Therapy) | Placebo + CBT (Prolonged Exposure Therapy) | Placebo + Supportive Counseling | Total
Number analyzed (Participants) | 42 | 40 | 40 | 43 | 165
Age, Continuous [Mean (Full Range); unit: years] | 44.9 [24 to 63] | 40.1 [19 to 64] | 44.7 [23 to 62] | 41.2 [24 to 58] | 42.7 [19 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 13 | 13 | 15 | 57
  Male | 26 | 27 | 27 | 28 | 108
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 21 | 30 | 28 | 26 | 105
  White | 19 | 9 | 8 | 14 | 50
  Hispanic | 2 | 1 | 3 | 1 | 7
  Native American | 0 | 0 | 0 | 1 | 1
  Other | 0 | 0 | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 40 | 40 | 43 | 165
Types of trauma [Count of Participants; unit: Participants]
  Sexual Assault | 11 | 12 | 11 | 8 | 42
  Physical Assault | 18 | 16 | 12 | 16 | 62
  Combat | 4 | 4 | 7 | 4 | 19
  Other | 9 | 8 | 10 | 15 | 42

OUTCOME MEASURES:

1. Primary Outcome: Posttraumatic Stress Disorder (PTSD) Symptom Scale - Interview (PSS-I-IV)
Description: The PSS-I-IV is a clinician-rated interview that evaluates PTSD symptoms on a frequency/severity scale corresponding to the DSM-IV symptom criteria. The measure has a total score range from 0 to 51, with higher scores indicating more severe PTSD symptoms.
Time Frame: Week 0 (Pretreatment), Week 24 (Posttreatment), Week 52 (Follow-up)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Naltrexone + Supportive Counseling | Naltrexone + CBT (Prolonged Exposure Therapy) | Placebo + CBT (Prolonged Exposure Therapy) | Placebo + Supportive Counseling
Number analyzed (Participants) | 42 | 40 | 40 | 43
units on a scale
  Pretreatment (Week 0) | 27.1 [24.7 to 30.8] | 30.3 [27.7 to 32.9] | 27.7 [24.7 to 30.8] | 27.5 [25.4 to 29.6]
  Posttreatmwent (Week 24) | 15.3 [12.2 to 18.3] | 12.2 [8.2 to 16.1] | 13.3 [9.3 to 17.3] | 15.5 [12.4 to 18.6]
  Follow-up (Week 52) | 10.9 [7.2 to 14.6] | 7.9 [4.1 to 11.8] | 10.8 [6.3 to 15.2] | 11.1 [8.2 to 14.1]

2. Primary Outcome: Drinking Timeline Follow-back Interview (TFBI)
Description: The TFBI is an interview that utilizes a calendar method to assess when and how much alcohol was consumed by the participant. At Week 0 (Pretreatment), Week 24 (Posttreatment), and Week 52 (Follow-up), alcohol consumed in the past 90 days was assessed. This measure was then used to calculate the percentage of days drinking in the past 90 days at each time point. Higher scores for percentage of days drinking indicate worse drinking outcomes.
Time Frame: Week 0 (Pretreatment), Week 24 (Posttreatment), Week 52 (Follow-up)
Measure: Mean (95% Confidence Interval); unit: percentage of days
Arm/Group | Naltrexone + Supportive Counseling | Naltrexone + CBT (Prolonged Exposure Therapy) | Placebo + CBT (Prolonged Exposure Therapy) | Placebo + Supportive Counseling
Number analyzed (Participants) | 42 | 40 | 40 | 43
percentage of days
  Pretreatment (Week 0) | 75.4 [67.1 to 83.5] | 71.2 [62.5 to 79.9] | 78.6 [71.4 to 85.6] | 74.1 [66.4 to 81.8]
  Posttreatmwent (Week 24) | 3.5 [0.1 to 6.8] | 7.3 [1.9 to 12.7] | 13.4 [5.5 to 21.1] | 13.2 [7.3 to 19.2]
  Follow-up (Week 52) | 21.5 [10.6 to 32.4] | 8.8 [3.3 to 14.3] | 18.9 [8.8 to 29.1] | 27.3 [14.7 to 40.0]

3. Secondary Outcome: Penn Alcohol Cravings Scale
Description: The Penn Alcohol Craving Scale is a 5-item self-report measure. It assesses alcohol craving during the prior week. Total scores on this measure range from 0 to 30, with higher scores indicating a higher level of craving.
Time Frame: Week 0 (Pretreatment), Week 24 (Posttreatment), Week 52 (Follow-up)
Measure: Mean (95% Confidence Interval); unit: percentage of days
Arm/Group | Naltrexone + Supportive Counseling | Naltrexone + CBT (Prolonged Exposure Therapy) | Placebo + CBT (Prolonged Exposure Therapy) | Placebo + Supportive Counseling
Number analyzed (Participants) | 42 | 40 | 40 | 43
percentage of days
  Pretreatment (Week 0) | 17.7 [15.3 to 20.0] | 17.9 [15.8 to 20.1] | 19.2 [16.3 to 22.1] | 18.7 [16.7 to 20.7]
  Posttreatmwent (Week 24) | 8.0 [6.0 to 10.0] | 5.1 [3.4 to 6.7] | 9.1 [6.1 to 12.2] | 10.3 [8.2 to 12.4]
  Follow-up (Week 52) | 7.4 [4.2 to 10.6] | 6.0 [4.0 to 8.1] | 6.9 [4.2 to 9.7] | 8.9 [6.4 to 11.4]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout time of participant enrollment and involvement in the study. Participant enrollment began on February 8, 2001 and ended on June 25, 2009. Data collection was completed on August 12, 2010. Therefore, adverse event data were collected for 9 years, 6 months.
Description: Please Note: None of the Serious Adverse events were determined to be related to the study.
Arm/Group | Naltrexone + Supportive Counseling | Naltrexone + CBT (Prolonged Exposure Therapy) | Placebo + CBT (Prolonged Exposure Therapy) | Placebo + Supportive Counseling
Serious Adverse Events (participants affected / at risk) | 3/42 | 2/40 | 4/40 | 3/43
Other Adverse Events (participants affected / at risk) | 21/42 | 21/40 | 22/40 | 18/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naltrexone + Supportive Counseling (N=42) | Naltrexone + CBT (Prolonged Exposure Therapy) (N=40) | Placebo + CBT (Prolonged Exposure Therapy) (N=40) | Placebo + Supportive Counseling (N=43)
Serious Suicidal Ideation (Psychiatric disorders) | 3 | 1 | 2 | 1
Serious Medical Illness (General disorders) | 0 | 1 | 1 | 1
Psychotic Symptoms (Psychiatric disorders) | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone + Supportive Counseling (N=42) | Naltrexone + CBT (Prolonged Exposure Therapy) (N=40) | Placebo + CBT (Prolonged Exposure Therapy) (N=40) | Placebo + Supportive Counseling (N=43)
Back Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (7)
Diarrhea (Renal and urinary disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Gastrointestinal Issues (Gastrointestinal disorders) | 3 (4) | 0 (0) | 1 (1) | 1 (1)
Changes to Vision (Eye disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
Toothache (General disorders) | 1 (3) | 0 (0) | 2 (2) | 2 (3)
Anxiety (General disorders) | 0 (0) | 3 (4) | 1 (2) | 0 (0)
Headache (General disorders) | 5 (8) | 9 (12) | 3 (5) | 3 (10)
Loose Stool (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (3)
Sedation (General disorders) | 2 (4) | 0 (0) | 1 (2) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 2 (3) | 1 (1) | 3 (6) | 0 (0)
Muscle Aches (General disorders) | 3 (3) | 0 (0) | 3 (4) | 0 (0)
Cold (Immune system disorders) | 5 (9) | 4 (4) | 5 (7) | 4 (4)
Nausea (Gastrointestinal disorders) | 10 (20) | 4 (5) | 7 (7) | 7 (11)
Dry Mouth (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Increased Bowel Movements (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (5) | 0 (0) | 0 (0)
Stomach Virus (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Increased Irritability (General disorders) | 2 (4) | 0 (0) | 2 (5) | 1 (1)
Fatigue (General disorders) | 4 (7) | 4 (5) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (3)
Dizziness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No